CLINICAL TRIAL: NCT03417115
Title: Treatment and Outcome of Patients With Breast Cancer: Clinical Research Platform for Real World Data
Brief Title: Breast Cancer Registry Platform
Acronym: OPAL
Status: Active, not recruiting | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-100361; Registerplattform OPAL (Other: iOMEDICO)
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Epidemiology; Registry; Health Services Research; Germany; Palliative Treatment; Adjuvant Treatment; Neoadjuvant Treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (6):
- Advanced breast cancer - Her2 positive: Patients with HER2-positive advanced breast cancer
- Advanced breast cancer - triple negative: Patients with triple negative advanced breast cancer
- Advanced breast cancer - HR positive, Her2 negative: Patients with HR positive, Her2 negative advanced breast cancer
- Early breast cancer - HER2 positive: Patients with HER2 positive early breast cancer
- Early breast cancer - triple negative: Patients with triple negative early breast cancer
- Early breast cancer - HR positive, HER2 negative: Patients with HR positive, HER2 negative early breast cancer

SUMMARY:
The purpose of the project is to set up a national, prospective, longitudinal, multicenter cohort study with associated satellites, a tumor registry platform, to document uniform data on characteristics, molecular diagnostics, treatment and course of disease, to collect patient-reported outcomes and to establish a decentralized biobank for patients with breast cancer in Germany.

DETAILED DESCRIPTION:
OPAL is a national, observational, prospective, longitudinal, multicenter cohort study (tumor registry platform) with the purpose to record information on the antineoplastic treatment of breast cancer in Germany. The registry will follow patients for up to five years. It will identify common therapeutic sequences and changes in the treatment of the disease. At inclusion, data in patient characteristics, comorbidities, tumor characteristics and previous treatments are collected. During the course of observation data on all systemic treatments, radiotherapies, surgeries, and outcome are documented.

Health-related quality of life in patients with breast cancer will be evaluated for up to five years.

ELIGIBILITY:
Inclusion Criteria:

EBC cohort:

* Female and male patients with early breast cancer (stage I-III defined as breast cancer that has not spread beyond the breast or the axillary lymph nodes)
* Patients at the start of their initial systemic treatment for EBC, i.e. at start of neoadjuvant treatment for patients receiving neoadjuvant thera-py or at start of adjuvant treatment if no neoadjuvant therapy is given. Treatment can be cytotoxic, endocrine, or targeted substances, what-ever was given first

ABC cohort:

* Female and male patients with advanced breast cancer (stage IV defined as synchronous or metachronous diagnosis of distant metastases at inclusion)
* Patients at the start of their initial first-line systemic treatment for ABC, which can be cytotoxic, endocrine or targeting a specific signaling pathway, whatever is given first

All cohorts:

* Written informed consent

  * Patients participating in the PRO module: signing of informed consent form and completion of baseline questionnaire before start of initial systemic treatment for EBC or systemic first-line treatment for ABC
  * Patients not participating in the PRO module: within six weeks after start of initial systemic treatment for EBC or systemic first-line treatment for ABC
* Age ≥ 18 years

Exclusion Criteria:

* Patients with prior systemic therapy (cytotoxic, endocrine, or targeted) for EBC or ABC
* Patients who do not receive any systemic therapy for EBC or ABC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female and male patients with breast cancer starting first systemic treatment for EBC or ABC.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-12-22 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Treatment reality | 5 years
  Description of treatment reality (Course of systemic treatments and sequential treatments) applied in German routine practice measured as the frequency of the various systemic treatments applied per line of therapy.

SECONDARY OUTCOMES:
Best Response | 5 years
  Documentation of response rates per line of treatment.
Progression-free survival | 5 years
  Documentation of progression-free survival per line of treatment.
Overall survival | 5 years
  Documentation of date of death.
Health-related quality of life (Patient-reported outcome) | 3.5 years
  EORTC QLQ-C30 core questionnaire and additional items.
Disease-free survival | 5 years
  Documentation of disease-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Marschner, MD, Study Chair — Praxis für interdisziplinäre Onkologie & Hämatologie
Locations (1):
- Multiple sites all over germany, Many Locations, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thill M, Zahn MO, Welt A, Stickeler E, Nusch A, Fietz T, Rauh J, Wetzel N, Kruggel L, Janicke M, Marschner N, Harbeck N, Wockel A, Decker T; OPAL study group. Treatment and outcome in metastatic lobular breast cancer in the prospective German research platform OPAL. Breast Cancer Res Treat. 2023 Apr;198(3):545-553. doi: 10.1007/s10549-023-06882-7. Epub 2023 Feb 18. PMID 36807725